CLINICAL TRIAL: NCT00909454
Title: V.I.P. Feasibility Study (Vitamin D Intake Project)
Brief Title: Vitamin D Supplement Study for Adolescents
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Yanbin Dong, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0901159
Record Dates: First submitted 2009-05-22; First posted 2009-05-28 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Vitamin D Deficiency; Overweight; Obesity
Keywords: Vitamin D deficiency; Adolescents; African Americans; Overweight; Obesity
MeSH Terms: conditions — Vitamin D Deficiency; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily 2000 IU vitamin D supplement (Experimental)
  Interventions: Dietary Supplement: 2000 IU Vitamin D3 daily supplement
- Daily Vitamin D supplement 400 IU (Active Comparator)
  Interventions: Dietary Supplement: 400 IU Vitamin D3 supplement

INTERVENTIONS:
Dietary Supplement: 2000 IU Vitamin D3 daily supplement — 2000 IU vitamin D3 supplement to be taken once daily over 4 months
  Other Names: NatureMade Maximum Strength D Vitamin 2000 IU List NO. 2516
  Arms: Daily 2000 IU vitamin D supplement
Dietary Supplement: 400 IU Vitamin D3 supplement — 400 IU Vitamin D3 supplement to be taken daily over 4 months
  Other Names: NatureMade D Vitamin 400 IU List No. 1688
  Arms: Daily Vitamin D supplement 400 IU

SUMMARY:
The purpose of this study is to determine if 14-19 year old African American adolescents are able to take a daily vitamin D supplement daily for about 4 months and how well a daily dose of 400 IU or 2000 IU vitamin D supplement raises their vitamin D blood level.

DETAILED DESCRIPTION:
To determine the feasibility of African American teenagers taking a daily vitamin D supplement over a 4 month period in terms of compliance and practical implementation.

To determine the differences in response in blood 25-OH D level between those randomly assigned to taking a 400 IU supplement versus 2000 IU per day and to determine if there are differences in blood 25-OH D level response depending on subject gender and overweight/obese versus healthy-weight status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy African American Adolescents

Exclusion Criteria:

* Hypertension
* Pregnancy
* Medications that affect study outcome measures
* Use of other vitamin and/or mineral supplement or herbal supplements
* Individuals of other races

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Plasma 25-OH D level | 3-4 months from baseline to post-testing

SECONDARY OUTCOMES:
Blood pressure | 3-4 months from baseline to post-testing

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute at Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Derived] Dong Y, Stallmann-Jorgensen IS, Pollock NK, Harris RA, Keeton D, Huang Y, Li K, Bassali R, Guo DH, Thomas J, Pierce GL, White J, Holick MF, Zhu H. A 16-week randomized clinical trial of 2000 international units daily vitamin D3 supplementation in black youth: 25-hydroxyvitamin D, adiposity, and arterial stiffness. J Clin Endocrinol Metab. 2010 Oct;95(10):4584-91. doi: 10.1210/jc.2010-0606. Epub 2010 Jul 21. PMID 20660028